CLINICAL TRIAL: NCT01538641
Title: Phase II Evaluation Of GROC (Gemcitabine- Rituximab-Oxaliplatin Combination) Given Every 14 Days For The Treatment Of Patients With Relapsed Or Refractory Aggressive Non-Hodgkin's Lymphoma
Brief Title: Phase II Evaluation of Gemcitabine- Rituximab-Oxaliplatin Combination (GROC) in Relapsed Aggressive Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Auxilio Mutuo Cancer Center (Other)
Responsible Party: Principal Investigator, Fernando Cabanillas, Hematology - Oncologist, Auxilio Mutuo Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCAM-03-01
Record Dates: First submitted 2012-02-21; First posted 2012-02-24 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Refractory Aggressive Non-Hodgkin's Lymphoma; Relapsing Aggressive Non-Hodgkin's Lymphoma
MeSH Terms: interventions — Rituximab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Rituximab, Gemcitabine, Oxaliplatin

INTERVENTIONS:
Drug: Rituximab, Gemcitabine, Oxaliplatin — Rituximab:375 mg/m2; on day 1 of each 14 days cycle. Gemcitabine:1,000 mg/m2 on day 2 of each 14 days cycle. Oxaliplatin:100 mg/m2; on day 2 of each 14 days cycle. Total number of cycles: 6 cycles.

SUMMARY:
Study Proposal:

Other drugs where synergy with Gemcitabine has been observed are Cisplatinum, Taxol, Taxotere, Etoposide and alkylating agents. However in view of Oxaliplatin's superior activity as a single agent against lymphoma, the combination of Gemcitabine with Oxaliplatin is more attractive and should be explored in this group of disorders. Based on these data and considering the advantage of its favorable toxicity profile, we propose a phase II study in patients with either refractory or relapsing aggressive non-Hodgkin's lymphomas including peripheral T-cell lymphomas which are known to have a poor outcome when compared with equivalent aggressive B-cell lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory or relapsed aggressive non-Hodgkin's Lymphoma. The definition of refractory includes patients who either did not respond to prior therapy or those whose best response was a PR after at least 4 courses of chemotherapy. Aggressive histologies include follicular large cell, diffuse large cell, peripheral T cell, transformed lymphomas, Lymphoblastic lymphomas, Burkitt and Burkitt like lymphomas.
* Histologic or cytological confirmation of refractory or relapsed aggressive non-Hodgkin's Lymphoma is desirable but not mandatory and will be left to the discretion of the investigator.
* Must have measurable or evaluable disease.
* No more than 4 previous regimens of chemotherapy will be allowed, including stem cell or bone marrow transplant.
* Patients must be more than 18 years old.
* No evidence of grade 3 or more neurosensory or neuromotor dysfunction (see appendix- toxicity criteria)
* Written Consent
* Those patients who have previously received a platinum or nucleoside analogue-containing regimen are eligible.
* Patients who are candidates for stem cell or marrow transplant will be included

Exclusion Criteria:

* Patients with a previous or concurrent history of cancer with the exception of: 1-treated carcinoma in situ of cervix or breast. 2- treated squamous or basal cell skin cancer, or 3- any other surgically cured malignancy from which the patient has been disease free for at least 5 years.
* HIV positive patients and those with Hepatitis B or C will be excluded from this protocol.
* Patients with severe neuropathy will be excluded.
* Chemotherapy or Radiotherapy within the previous 3 weeks prior to entering study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2003-10; Primary Completion 2007-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The response rate of the combination of Gemcitabine-Oxaliplatin-Rituximab. | 5 years